CLINICAL TRIAL: NCT01671826
Title: Prospective, Observational, Multicenter Trial Evaluating Autologous Stem Cell Transplantation for Myeloma Patients Over the Age of 65
Brief Title: Autologous Stem Cell Transplantation for Myeloma Patients Over 65 Years
Acronym: LATMM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: LGT-2012
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Newly Diagnosed Myeloma Patient Above 65 Years Old
Keywords: Multiple Myeloma; Autologous Stem Cell Transplantation; Elderly Patients
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- above 65 years old

SUMMARY:
Autologous stem cell transplantation remains the gold standard of treatment for newly diagnosed patients under the age of 65. Even though it is also regularly performed above the age of 65, there are very few data in this patient population. The investigators will capture safety and efficacy data in that setting.

DETAILED DESCRIPTION:
Newly diagnosed myeloma patients above the age of 65 years will be treated the following way: Bortezomib (Velcade®) based induction treatment (either Velcade Dexamethasone, Velcade Thalidomide Dexamethasone (VTD) or Velcade Cyclophosphamide Dexamethasone (VCD)). After the induction phase, for patients at least in partial remission, a collection of peripheral blood stem cells (PBSC) is done according to each center practice. High dose melphalan (140 mg/m2) followed by PBSC autologous transplantation is then performed. Three months post transplant, 2-3 cycles (similar to the initial induction phase) of consolidation are allowed.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed MM,
* age over 65,
* measurable disease

Exclusion Criteria:

* Patients less than 65 and/or not proceeding to autologous PBSC transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed myeloma patients over 65 years of age and a measurable disease.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free survival | 2 years

SECONDARY OUTCOMES:
Response | after induction, 3 months post transplant, 2 months post consolidation
Time To Progression | 2 years
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Garderet, MD, Principal Investigator — Assistance Publique
Locations (6):
- France (6):
  - CHU, Dijon
  - CHU, Lille
  - CHU, Lyon
  - Institut Paoli Calmette, Marseille
  - CHU, Nantes
  - Hôpital Saint Antoine, Paris

REFERENCES:
- [Derived] Garderet L, Beohou E, Caillot D, Stoppa AM, Touzeau C, Chretien ML, Karlin L, Moreau P, Fontan J, Blaise D, Polge E, Gueye MS, Ikhlef S, Marjanovic Z, Labopin M, Mohty M. Upfront autologous stem cell transplantation for newly diagnosed elderly multiple myeloma patients: a prospective multicenter study. Haematologica. 2016 Nov;101(11):1390-1397. doi: 10.3324/haematol.2016.150334. Epub 2016 Sep 9. PMID 27612987